CLINICAL TRIAL: NCT00823407
Title: Clinical Pharmacology of MDA [3,4-methylenedioxyamphetamine]
Acronym: MDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, John Mendelson, MD, Senior Scientist, California Pacific Medical Center Research Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 27.112; IND# 79,632; 5R01DA016776 (NIH); CHR# H6637-31759-01; IRB# 27.112; RAP-C# 0740
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: MDA; MDMA; Ecstasy; entactogen; pharmacokinetics; pharmacodynamics; Pharmacokinetics and pharmacodynamics of MDA studies in healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDA (Other)
  Interventions: Drug: MDA; Drug: Placebo

INTERVENTIONS:
Drug: MDA — subjects will receive a single oral dose of MDA 98mg/70kg body weight
Drug: Placebo — Subjects will receive a single oral dose of placebo

SUMMARY:
The purpose of this study is to investigate the pharmacological and cognitive effects of MDA in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females age 18-50
* Fluent English speaker
* Willing and able to give written consent

Exclusion Criteria:

* Body mass index > 30 or < 18
* Pregnancy or lactation

FOR MORE DETAILS CONTACT THE RESEARCH CLINIC.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
MDA will be metabolized to hydroxyamphetamine (HMA) and dihydroxyamphetamine (DHA) and will produce dose-dependent increases in neuroendocrine measures. | 0-48 hours post dose

SECONDARY OUTCOMES:
MDA will produce dose-dependent increases in self-report entactogen-like and stimulant like measures. | 0-48 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: John E Mendelson, MD, Principal Investigator — CPMC Research Institute
Locations (1):
- CPMC Addiction & Pharmacology Research Laboratory (APRL), San Francisco, California, United States

REFERENCES:
- [Result] Baggott MJ, Siegrist JD, Galloway GP, Robertson LC, Coyle JR, Mendelson JE. Investigating the mechanisms of hallucinogen-induced visions using 3,4-methylenedioxyamphetamine (MDA): a randomized controlled trial in humans. PLoS One. 2010 Dec 2;5(12):e14074. doi: 10.1371/journal.pone.0014074. PMID 21152030
- See also: Addiction & Pharmacology Research Laboratory webpage — http://www.cpmc.org/professionals/research/programs/addiction.html
- See also: PLoS ONE — http://www.plosone.org/article/info%3Adoi%2F10.1371%2Fjournal.pone.0014074